CLINICAL TRIAL: NCT03887793
Title: Quality Improvement Strategies to Increase Human Papillomavirus (HPV) Vaccination in Integrated Healthcare Delivery Systems
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate recruitment of study clinics
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); American Cancer Society, Inc. (Other); Wisconsin Department of Health and Family Services (Other Government); New York State Department of Health (Other Government); Association of Immunization Managers (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-0146b; 1U01IP001073-01 (NIH)
Record Dates: First submitted 2019-02-26; First posted 2019-03-25 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Human Papillomavirus Infection
Keywords: quality improvement; HPV vaccine; integrated healthcare delivery systems
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VACs intervention (Experimental): Integrated healthcare delivery systems randomly assigned to this arm will participate in the Vaccinate Adolescents against Cancers (VACs) model for HPV vaccine QI. Specific QI activities will be chosen by healthcare system leadership and healthcare providers on the systems' QI teams.
  Interventions: Other: VACs
- Wait list control (No Intervention): Integrated healthcare delivery systems randomly assigned to this arm will be placed on a waiting list to receive the intervention after the conclusion of the study period.

INTERVENTIONS:
Other: VACs — The VACs (Vaccinate Adolescents against Cancer) model for HPV vaccine quality improvement is a strategy developed by the American Cancer Society to improve HPV vaccination coverage in large integrated health care delivery systems. It includes the development of a quality improvement (QI) action plan, the formation of a QI team of health care providers, education for the QI team about HPV-related disease burden and vaccine efficacy, HPV vaccine coverage assessments at several time points that are shared with individual clinics within the health are system, and the adoption of specific QI strategies by participating clinics in the health care system.
  Arms: VACs intervention

SUMMARY:
HPV vaccination coverage is at lower levels than the national goal. This study will evaluate the effectiveness of quality improvement strategies for increasing HPV vaccination coverage among adolescent within the context of large integrated health care delivery systems.

DETAILED DESCRIPTION:
The University of North Carolina (UNC) will evaluate the impact of a quality improvement (QI) model for increasing HPV vaccination coverage among adolescents in primary care settings. UNC will partner with the American Cancer Society (ACS) to evaluate the effectiveness of their Vaccinate Adolescents against Cancer (VACs) model for HPV vaccine QI within the context of integrated healthcare delivery systems (IDSs). The VACs model includes the development of a QI action plan and a QI team. The QI team is made up of health care providers from participating clinics within the IDSs. The team then helps implement specific QI activities in participating primary care clinics. The model also includes vaccination coverage assessments in participating clinics at multiple time points to assess the impact of QI activities. Specific QI activities that will be offered to participating clinics will be chosen from a menu of options that will include the Center for Disease Control and Prevention's AFIX model and physician-to-physician engagement. AFIX (Assessment, Feedback, Incentives and eXchange) consists of brief quality improvement consultations that immunization specialists from state health departments deliver to vaccine providers in primary care settings. Using immunization registry data, the specialist evaluates the clinic's vaccination coverage and delivers education on best practices to improve coverage. Physician-to-physician (P2P) engagement consists of an in-depth training about how to make strong and effective HPV vaccination recommendations to primary care providers. The investigators will compare changes in HPV vaccination coverage between the quality improvement arm or wait list control arm.

ELIGIBILITY:
Inclusion Criteria:

* Integrated healthcare delivery systems headquartered in New York State or Wisconsin with at least 4 pediatric or internal medicine practices within the system.
* All clinics within the integrated healthcare delivery system must participate in the state immunization registry.

Exclusion Criteria:

* Integrated healthcare delivery systems headquartered outside of New York State or Wisconsin.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
HPV vaccination (≥1 dose), 11-12 year olds at 6 months | Six months
  Coverage change from baseline to 6 months in HPV vaccine initiation (≥1 dose), among 11- to 12- year old patients, as measured by states' immunization information system (IIS) records

SECONDARY OUTCOMES:
HPV vaccination (≥1 dose), 11-12 year olds at 6 months by state | Six months
  Coverage change from baseline to 6 months in HPV vaccine initiation (≥1 dose), among 11- to 12- year-old patients, as measured by states' IIS records, stratifying by state (NY or WI)
HPV vaccination (completion according to the Advisory Committee on Immunization Practices (ACIP) guidelines), 11-12 year olds at six months | Six months
  Coverage change from baseline to six months in HPV vaccine completion, among 11- to 12- year-old patients, as measured by states' IIS records
HPV vaccination (completion according to the Advisory Committee on Immunization Practices (ACIP) guidelines), 11-12 year olds at six months by state | Six months
  Coverage change from baseline to six months in HPV vaccine completion, among 11- to 12- year-old patients by state (NY or WI), as measured by states' IIS records
HPV vaccination (≥1 dose), 13-17 year olds at six months | Six months
  Coverage change from baseline to six months in HPV vaccine initiation (≥1 dose), among 13- to 17- year-old patients, as measured by states' IIS records
HPV vaccination (completion according to ACIP guidelines), 13-17 year olds at six months | Six months
  Coverage change from baseline to six months in HPV vaccine completion, among 13- to 17- year-old patients, as measured by states' IIS records

CONTACTS AND LOCATIONS:
Overall Officials: Noel T Brewer, PhD, Principal Investigator — University of North Carolina; Melissa B Gilkey, PhD, Principal Investigator — University of North Carolina
Locations (2):
- United States (2):
  - New York State Department of Health, Albany, New York
  - Wisconsin Department of Health Services, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No